CLINICAL TRIAL: NCT04615702
Title: Evidence Based Management of Acute Biliary Pancreatitis
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, yasmine Hany Hegab, principal investigator, Zagazig University
Other Study IDs: acute panreatitis guidelines
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis guidelines; acute biliary pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ultrasonography; Endosonography; Ringer's Lactate; Anti-Inflammatory Agents, Non-Steroidal; Diclofenac; Acetaminophen; Opiate Alkaloids; Meperidine; Quinolones; Metronidazole; Ciprofloxacin; Carbapenems; Imipenem; Fresubin; Enteral Nutrition; Apoptosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- application of recent guidelines in the management of acute biliary pancreatitis: all patients subjected to the following: Confirmation of the diagnosis of acute pancreatitis, Diagnosis of the cause either biliary or not, Severity scoring and Evidence based management regarding Initial management, Intervention as indicated, Prevention of recurrence and Follow up
  Interventions: Diagnostic Test: serum lipase or amylase; Device: ultrasound; Device: CT; Diagnostic Test: Liver enzymes (Bilirubin, alanine transferase (ALT), aspartate aminotransferase, (AST) and alkaline phosphatase). Calcium. Triglycerides.; Device: EUS /Secretin-stimulated magnetic resonance cholangiopancreatography (MRCP); Drug: Ringer lactate; Combination Product: NSAID / paracetamol +/- opiates+/- epidural analgesia; Combination Product: Quinolones + Metronidazole /Carbapenems ± Metronidazole; Dietary Supplement: Fresubin 2Kcal fiber drink; Device: nasogastric tube; Procedure: retroperitoneal necrosectomy; Procedure: open necrosectomy; Procedure: Endoscopic transmural cystogastrostomy; Procedure: open cystogastrostomy; Procedure: percutaneous catheter drainage (PCD) for infected necrosis; Procedure: Endoscopic ultrasound (EUS) guided aspiration for infected necrosis

INTERVENTIONS:
Diagnostic Test: serum lipase or amylase — Laboratory ( elevated serum lipase or amylase at least 3 times above the normal limits) is helpful in diagnosis
  Acute pancreatitis is diagnosed when two of three criteria are present including:
  1. Clinically (abdominal pain consistent with acute pancreatitis),
  2. Laboratory ( elevated serum lipase or amylase at least 3 times above the normal limits)
  3. Imaging criteria of acute pancreatitis
Device: ultrasound — helpful in diagnosis of acute pancreatitis and its etiology (Gallstones)
Device: CT — helpful in diagnosis of acute pancreatitis and its etiology . assist in detection of type and severity of acute pancreatitis
Diagnostic Test: Liver enzymes (Bilirubin, alanine transferase (ALT), aspartate aminotransferase, (AST) and alkaline phosphatase). Calcium. Triglycerides. — help in diagnosis of the etiology of acute pancreatitis elevated Bilirubin, ALT, AST and alkaline phosphatase suggest biliary pancreatitis
Device: EUS /Secretin-stimulated magnetic resonance cholangiopancreatography (MRCP) — helpful in idiopathic acute pancreatitis diagnosis
Drug: Ringer lactate — The initial infusion rate for mild cases :
  * For patients without dehydration is (130-150mL/h).
  * In case of dehydration: (150-600mL/h) with close monitoring of patients with comorbidities such as cardiac problems or renal failure to avoid volume overload.
  The initial infusion rate for both severe cases :
  * For patients without dehydration is (130-150mL/h).
  * In case of dehydration/ shock: (150-600mL/h) with close monitoring of patients with comorbidities such as cardiac problems or renal failure to avoid volume overload d. The target
  * A mean arterial pressure of 65mmHg or more,
  * Urine output of 0.5mL/kg per hour or more When these parameters achieved, the infusion rate decreased to the level that maintain these parameters.
  Other Names: hartmann's solution
Combination Product: NSAID / paracetamol +/- opiates+/- epidural analgesia — Pain control (Modified World Health organization (WHO) analgesia ladder) Step1: NSAID / paracetamol Paracetamol 1gm IV infusion /8h + Diclofenac sodium 75mg /12h.
  Step 2: Opiates +/- NSAID/ paracetamol Pethidine 25 mg IV/4h
  Step 3: Interventional treatment (epidural analgesia) +/- opiates +/- NSAID/ paracetamol In case of severe pain not responding to the above analgesia
  Other Names: NSAID (Diclofenac sodium) paracetamol (perfalgan drip) Opiates (Pethidine)
Combination Product: Quinolones + Metronidazole /Carbapenems ± Metronidazole — * Mild attack: no antibiotic prophylaxis administered.
  * Severe attack:
  * Timing: Antibiotic prophylaxis administered to cases presented early within 72 hrs of disease onset.
  * Duration: Not more than 2 weeks
  * Antibiotics given:
    * Quinolones + Metronidazole ( the 1st choice in ward) Ciprofloxacin 400mg IV /12 h + metronidazole 500mg IV/8h
    * Carbapenems ± Metronidazole (the 1st choice in ICU patients and in case of sensitivity to quinolones) Imipenem .5gm IV/6h + metronidazole 500mg IV/8h
      b. Therapeutic (in cases with pancreatic or extrapancreatic infections)
    * In case of pancreatic infection, Carbapenems ± metronidazole were given.
  Other Names: Quinolones (ciprofloxacin) Metronidazole (flagyl) Carbapenems (Imipenem)
Dietary Supplement: Fresubin 2Kcal fiber drink — Severe cases Timing: Within at least 48 hrs of admission provided that there are no intestinal complications.
  Route: Nasogastric tube Nutrients: Polymeric feeding formula
  * Nutrient: Fresubin 2Kcal fiber drink 200ml (2Kcal/ml)
  * Total caloric requirements ꞊ body weight (kg) X 30Kcal/day Pattern : Continuous infusion
  * The nutrition started with small amount and increased gradually over 16hrs
  * Infusion rate ꞊ Total caloric requirements / 16hrs
  Other Names: polymeric feeding formula
Device: nasogastric tube — in case of ileus or vomiting
Procedure: retroperitoneal necrosectomy — * General anesthesia , Supine position with 30 degree tilt towards the right side
  * A left subcostal 5 cm incision is performed one finger below the left costal margin over the midaxillary line and the muscles were divided sequentially
  * Then, aspiration is done from the possible collection.
  * After confirmation that it was the site of the collection, the fibrotic thick wall was opened by a scissor, as the collection is opened, pus drained spontaneously.
  * At first, a wide suction was introduced in the cavity and the friable loose necrotic tissue was aspirated. Then, a circuit of flushing saline was created in the residual cavity by injection of saline through the previously placed PCD followed by aspiration of the saline and detached loose necrotic tissue fragments by the wide suction tube
  * After completion of the procedure, large bore surgical drain was placed into the collection. The fascia was closed over the drains. The skin closed by interrupted sutures
Procedure: open necrosectomy — Open necrosectomy was done after failure of the minimally invasive techniques. The procedure was done under general anesthesia under the coverage of Tienam (.5gm/6h IV) following the results of culture and sensitivity of the percutaneous drain effluent Surgical exploration of the peritoneal cavity was done through midline exploratory incision, there were 2 large pus collections extending from the Rt. and Lt. Lumber regions deep down into the pelvis, the intervening septa were divided and the pus was aspirated by a wide suction drain.
  The lesser sac was opened and necrosectomy was done The previously placed PCD repositioned in the site of necrosectomy as a port for continuous irrigation while a wide tube drain was placed in the lesser sac for drainage. Another 2 tube drains were placed in the pelvis.
Procedure: Endoscopic transmural cystogastrostomy — for pancreatic pseudocyst Antibiotic prophylaxis with Ciprofloxacin 400mg IV /12 hour was administered before the procedure and continued for 5 days after the procedure At first the cyst morphology was evaluated by EUS and color Doppler ultrasound is used to identify nearby vessels The puncture was performed using a 19-gauge needle, which was introduced into the pseudocyst via a therapeutic linear array echoendoscope. Then, a 0.035-inch guidewire was introduced through the needle and coiled within the pseudocyst under fluoroscopic guidance.
  The needle was removed and a 10F cystotome was advanced over the guidewire and the tract was dilated by the cystotome, after dilatation, a 10F double-pigtail stent was placed and a sample of the aspirate is sent for chemical and microbiological analysis
Procedure: open cystogastrostomy — for pancreatic pseudocyst general anesthesia, 1 gm of cefotax was given IV at the induction of anaesthesia, supine position over the operating table A transverse supraumbilical incision was performed. A 5 cm horizontal anterior gastrotomy was performed (Image 23a). Hemostasis of the submucosal vessels was performed before the incision of the gastric mucosa.
  First, the cyst was punctured followed by an incision of 5 cm at the posterior gastric wall. Aspiration of the cyst content was done for chemical and microbiological analysis The wall of the pseudocyst is hemmed to the gastric wall with continuous sutures made of a vicryl 2/0 alongside the entire circumference of the orifice Nasogastric tube was placed in the stomach. The procedure was completed by suturing the anterior gastrotomy with a vicryl 2/0 continous sutures in 2 layers A tube drain was inserted at the pelvis with closure of the abdominal wound in a standard way.
Procedure: percutaneous catheter drainage (PCD) for infected necrosis — PCD
  * The percutaneous drainage catheter placed through peritoneal approach under US guidance, the drain size was 12 F.
  * After placement of the percutaneous catheter, aspirate was sent for microbiological assessment
  * The PCD was flushed with 50 ml saline, three times daily to keep the drain open and improve lavage of the collection
Procedure: Endoscopic ultrasound (EUS) guided aspiration for infected necrosis — endoscopic approach it was done to one patient in the form of EUS guided aspiration of pus in a case with infected necrosis followed by percutaneous US guided aspiration of the residual

SUMMARY:
This study aims to assess the outcome of standardized evidence-based care to all patients with acute biliary pancreatitis treated at surgery department, Zagazig University hospitals during the period from may, 2017 to may 2019.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is one of the most important gastrointestinal disorders causing emotional and physical human burden . The annual incidence worldwide for AP is 4.9-73.4 cases per 100,000 people and the overall mortality rate is 4 to 8%, which increases to 33% in patients with infected necrosis. AP is diagnosed when two of three criteria are fulfilled: typical abdominal pain of AP, more than three times elevated serum amylase/lipase level and signs of AP on imaging.

It is necessary to clarify the etiology of AP promptly. The diagnosis of gallstones, as the leading cause for AP, should have the top priority as that will direct the treatment policy. Long standing alcohol consumption and gallstones disease incriminated in the majority of cases with AP. Small common bile duct stones, in particular, are the cause of AP in approximately 32 to 40% of cases. In 10-30% of cases, the cause is unknown, so studies have suggested that up to 70% of cases of idiopathic pancreatitis are secondary to biliary microlithiasis.

The pathogenesis of biliary AP has been intensively investigated. Many theories explain how gallstones can trigger AP. The predominant theories include common pathway theory and gallstone migration theory. In general, AP occurs when intracellular protective mechanisms fail to prevent trypsinogen activation or reduce trypsin activity.

It is important that management of such potentially life threatening condition to be guided by an evidence-based approach. After comparing the Japanese (JPN) Guidelines 2015 and its former edition 2010 with the other two guidelines, International Association of Pancreatology/American Pancreas Association guidelines (IAP/APA), 2013 and American College of Gastroenterology (ACG), 2013, the JPN Guidelines, 2015 proved to be the highest quality regarding its systematic literature review prepared by the meta-analysis team, including the grading of recommendations and providing pancreatitis bundles.

ELIGIBILITY:
Inclusion Criteria:

* all cases with acute biliary pancreatitis

Exclusion Criteria:

* all cases with non biliary pancreatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases with acute biliary pancreatitis admitted to surgery department in the study period were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
success rate of minimally invasive techniques (percutaneaous catheter drainage, endoscopic approach and retroperitoneal approach) in cases with infected walled off necrosis | immediately following intervention to 6 weeks following intervention
  Data were tabulated and statistically analyzed in terms of percentages Success of the intervention means patient condition improves [clinical (vital signs) , laboratory (CBC, kidney and liver function tests) and radiological improvement (no residual collection in CT)] and that there is no need for further intervention to control the disease till patient discharge
rate of complications of minimally invasive techniques used in the management of cases with infected walled off necrosis including bleeding, fistula, wound infection, incisional hernia | up to 6 months following intervention
  Data were tabulated and statistically analyzed in terms of percentages
Mortality rate of acute biliary pancreatitis in the study period | from admission to 6 months following admission
  Data were tabulated and statistically analyzed in terms of percentages
length of hospital stay of mild and severe cases with acute biliary pancreatitis | up to 6 months
  Data were tabulated and statistically analyzed in terms of frequencies length of hospital stay in days

SECONDARY OUTCOMES:
age of cases with acute biliary pancreatitis in Sharqia in years | at admission
  Data were tabulated and statistically analyzed in terms of mean
Sex of cases with acute biliary pancreatitis in Sharqia (Males and females) | at admission
  Data were tabulated and statistically analyzed in terms of percentages

CONTACTS AND LOCATIONS:
Overall Officials: yasmine Hegab, Principal Investigator — zagazig university faculty of human medicine
Locations (1):
- Zagazig University Faculty of Human Medicine, Zagazig, Egypt

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Result] Isaji S, Takada T, Mayumi T, Yoshida M, Wada K, Yokoe M, Itoi T, Gabata T. Revised Japanese guidelines for the management of acute pancreatitis 2015: revised concepts and updated points. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):433-45. doi: 10.1002/jhbp.260. PMID 25904407
- [Result] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Result] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878